CLINICAL TRIAL: NCT02886559
Title: Chidamide Plus DCAG for Relapsed/Refractory AML
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Navy General Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Li Yu, Professor, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CN301-XYK-003
Record Dates: First submitted 2016-08-29; First posted 2016-09-01 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2016-09

CONDITIONS: AML; Relapse
Keywords: demethylating agent; chidamide
MeSH Terms: conditions — Recurrence | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DCCAG (Experimental): Chidamide 30mg twice for one week decitabine 20mg/m^2 for 5 days
  Interventions: Drug: Chidamide plus DCAG regimen

INTERVENTIONS:
Drug: Chidamide plus DCAG regimen — chidamide, decitabine, aclarubicin, cytarabine and G-CSF
  Other Names: DCCAG regimen

SUMMARY:
Despite advances in understanding the complexities of acute myeloid leukaemia (AML), the treatment of refractory or relapsed AML (rrAML) remains a daunting clinical challenge.The investigators designed a new regimen, including chidamide, decitabine, aclarubincin, cytarabine and G-CSF, to treat rrAML.

ELIGIBILITY:
Inclusion Criteria:

* Men and women whose age more than 18 and less than 59；
* Patients diagnosed as AML according to the 2008 WHO (WHO) myeloid malignant disease diagnosis standard;
* Patients who relapsed after remission or who can not achieve remission after at least two cycle of systemic therapy (including chemotherapy, hematopoietic stem cell transplantation, etc.);
* ECOG performance status 0-3;
* Expected survival time ˃ 3 months;
* Patients without serious hearts, lung, liver, kidney disease;
* Patients have not received radiotherapy, chemotherapy, targeted therapy or hematopoietic stem cell transplantation and other treatment within 4 weeks prior to the enrollment;
* Patients are able to understand and willing to sign informed consent.

Exclusion Criteria:

* Patients who allergy to the study drug or the drug with similar chemical structure;;
* Pregnancy, lactation women and women of childbearing age who do not want to practice effective methods of contraception;
* Active infection;
* Drug abuse, long-term alcohol abuse so as to affect the results of the evaluation of patients;
* Patients with mental disorders or other conditions can not obtain informed consent, can not meet the requirements of the study treatment and procedures;
* Patients have clinical significant QTc interval prolongation history (male > 450ms. Female >470ms), ventricular heart had tachycardia (VT) and atrial fibrillation (AF), II degree heart block, myocardial infarction attack (MI) within 1 year prior to the enrollment, congestive heart failure (CHF), patients of coronary heart disease who have clinical symptoms and need drug treatment.
* Cardiac ultrasound showed that the diastolic pericardial fluid dark area width ˃ 10mm;
* Patients have received organ transplantation;
* Active bleeding
* Patients have new thrombosis, embolism, cerebral hemorrhage and other diseases or medical history of patients within 1 year prior to enrollment;
* The main organs of the surgery is less than 6 weeks;
* Bone marrow hyperplasia and WBC <2.0 * 10^9/L;
* Liver function abnormalities (total bilirubin > 1.5 times of upper limit of normal range , ALT / AST > 2.5 times of the upper limit of normal range or patients with liver involvement whose ALT / AST > 1.5 times of upper limit of normal range), renal anomalies (serum creatinine > 1.5 times of upper limit of normal value );
* Not suitable for the study according to investigator's assessment.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
overall response rate | 3 months

SECONDARY OUTCOMES:
overall survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Li Yu, MD. Ph.D, Study Chair — Chinese PLA General Hospital; Li-Xin Wang, MD. Ph.D., Principal Investigator — Navy General Hospital, Beijing, China
Locations (1):
- China PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Wang L, Luo J, Chen G, Fang M, Wei X, Li Y, Liu Z, Zhang Y, Gao S, Shen J, Wang X, Gao X, Zhou W, Ma Y, Liu H, Li X, Yang L, Sun K, Yu L. Chidamide, decitabine, cytarabine, aclarubicin, and granulocyte colony-stimulating factor (CDCAG) in patients with relapsed/refractory acute myeloid leukemia: a single-arm, phase 1/2 study. Clin Epigenetics. 2020 Sep 1;12(1):132. doi: 10.1186/s13148-020-00923-4. PMID 32873343